CLINICAL TRIAL: NCT03239314
Title: The Effect of Adding Dexamethasone to Bupivacaine in Ultrasound Guided Adductor Canal Block for Postoperative Analgesia Following Knee Arthroscopic Anterior Cruciate Ligament Reconstruction
Brief Title: Analgesic Effect of Adductor Canal Block With and Without Dexamethasone for Knee Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed galal aly, Assistant Professor of Anesthesia, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17100210
Record Dates: First submitted 2017-07-24; First posted 2017-08-04 (Actual); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Postoperative Analgesia
MeSH Terms: interventions — Saline Solution; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group I (Active Comparator): Group I (MS): received single shot 20 ml 0.5% isobaric bupivacaine + 2.0 ml normal saline solution injected into the adductor canal preoperatively.
  Interventions: Drug: Saline Solution
- group II (Active Comparator): Group II (MD): received 20 ml 0.5% isobaric bupivacaine + 8.0 mg dexamethasone (2.0 ml) injected into adductor canal preoperatively.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Saline Solution — Injected in the adductor canal
  Other Names: Normal Saline Solution
  Arms: group I
Drug: Dexamethasone — Injected in the adductor canal
  Other Names: Decadron
  Arms: group II

SUMMARY:
The purpose of this study was to evaluate the efficacy of ultra-sound guided adductor canal block with and without dexamethasone when added to bupivacaine on the duration of postoperative analgesia in patients undergoing arthroscopic anterior cruciate ligament reconstruction surgery using Numeric Rating Score (NRS).

DETAILED DESCRIPTION:
Adductor canal block was done by Ultra-sound. After confirmation of the block and exclusion of any signs of toxicity or nerve injury, the patients operations were done under spinal anesthesia. Patients were allocated into one of 2 groups (30 patients per group).

I. Group I: the patients received a single-shot of 20 ml plain bupivacaine (0.5%) +2 ml normal saline.

ii.Group II: the patients received 20ml plain bupivacaine (0.5%) + 8 mg dexamethasone (2ml).

Postoperative pain were assessed by Numeric Rating Scale (N.R.S) every 6 h post-operatively for 24 h.

Whenever, the NRS Score was ≥4 or the patient requested pain medication, analgesia was provided by ketorolac 30 mg amp IV, then morphine 1mg ̸ kg slowly IV as a rescue analgesia. Time to first request for analgesia & total dose of rescue analgesia were be recorded.

10. Satisfaction score will be measured on a linear numerical scale; ranging from 0 = complete dissatisfaction to 10 = complete satisfaction. Any post-operative side effects, like nausea, vomiting, bradycardia, hypotension will be also documented. The time to first analgesic requirement will be recorded, and the cumulative, post-operative opioid consumption in 24 h post-operatively will be recorded. Assessment of Quadriceps Strength at preoperative, 6, 12, 18, and 24 h postoperative from zero to 5.

ELIGIBILITY:
Inclusion Criteria:

* Adult ASA I-II Arthroscopic anterior cruciate ligament reconstruction

Exclusion Criteria:

* patient refusal
* drug allergy
* failed procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07-22 (Actual)

PRIMARY OUTCOMES:
duration of postoperative analgesia | One day postoperative
  assessed by pain score

SECONDARY OUTCOMES:
postoperative analgesic consumption | One day postoperative
  postoperative opioid consumption

REFERENCES:
- [Result] Rasouli MR, Viscusi ER. Adductor Canal Block for Knee Surgeries: An Emerging Analgesic Technique. Arch Bone Jt Surg. 2017 May;5(3):131-132. No abstract available. PMID 28656158
- [Derived] Ibrahim AS, Aly MG, Farrag WS, Gad El-Rab NA, Said HG, Saad AH. Ultrasound-guided adductor canal block after arthroscopic anterior cruciate ligament reconstruction: Effect of adding dexamethasone to bupivacaine, a randomized controlled trial. Eur J Pain. 2019 Jan;23(1):135-141. doi: 10.1002/ejp.1292. Epub 2018 Aug 6. PMID 30066465